CLINICAL TRIAL: NCT04178434
Title: E-health Treatment of Stress and Anxiety in Stockholm Myocardial Infarction With Non-obstructive Coronaries Study
Brief Title: Internet-based Treatment of Stress and Anxiety in Myocardial Infarction With Non-obstructive Coronary Arteries
Acronym: e-SMINC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Per Tornvall (Other)
Collaborators: Uppsala University (Other); Mid Sweden University (Other)
Responsible Party: Sponsor-Investigator, Per Tornvall, Professor, Karolinska Institutet
Organization: Karolinska Institutet (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20191111
Record Dates: First submitted 2019-11-11; First posted 2019-11-26 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Myocardial Infarction
Keywords: Myocardial infarction; Non-obstructive coronary arteries; Takotsubo syndrome
MeSH Terms: conditions — Myocardial Infarction; Takotsubo Cardiomyopathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Internet-based CBT intervention (Active Comparator): A nine step internet-based intervention with focus on stress and anxiety
  Interventions: Behavioral: Internet-based CBT intervention
- Treatment as usual (No Intervention): Regular follow-up with two doctor and one nurse appointment

INTERVENTIONS:
Behavioral: Internet-based CBT intervention — A nine step intervention including internet-based feedback by psychologists
  Arms: Internet-based CBT intervention

SUMMARY:
Patient with myocardial infarction with non-obstructive coronary arteries and takotsubo syndrome often have high levels of stress and anxiety. At present there are no treatment alternatives in this group of patients. Previously, cognitive behavioral therapy (CBT), primarily aiming at relieving stress, has been shown to decrease morbidity in patient with myocardial infarction with obstructive coronary arteries. The present open randomized study aims to decrease stress and anxiety in patients with myocardial infarction with non-obstructive coronary arteries and takotsubo syndrome by an internet-based CBT focusing on stress and anxiety.

ELIGIBILITY:
Inclusion Criteria:

* a suspected diagnosis of MINOCA or takotsubo syndrome with coronary angiography without diameter stenosis ≥50%
* age 35-80 years
* admission-ECG with sinus rhythm
* PSS-14 ≥ 25 and/or HADS-A ≥ 8 during admission
* reading and writing proficiency in Swedish
* computer/Internet access and literacy

Exclusion Criteria:

* strong clinical suspicion of myocarditis
* spontaneous coronary artery dissection
* acute pulmonary embolism
* acute myocardial infarction type 2
* cardiomyopathy other than takotsubo syndrome
* a previous myocardial infarction due to CAD
* expected poor compliance to behavioural therapy
* not likely to survive > one year due to for example cancer

Ages: 35 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2021-11-11 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Self-rated stress as determined by Perceived Stress Scale 14 (PSS-14) | 12-14 weeks after the acute event
  Normalisation of PSS-14 (<25 on a scale 0-56 with high numbers indicating increased stress)
Self-rated anxiety as determined by Hospital Anxiety and Depression Scale (HADS) | 12-14 weeks after the acute event
  Normalisation of HADS-A (<8 on a scale 0-21 with high numbers indicating increased anxiety)

SECONDARY OUTCOMES:
Self-rated stress as determined by Perceived Stress Scale 14 (PSS-14) | 10, 20 and 50 weeks after randomisation
  PSS-14 (<25 on a scale 0-56 with high numbers indicating increased stress)
Self-rated anxiety as determined by Hospital Anxiety and Depression Scale (HADS) | 10, 20 and 50 weeks after randomisation
  HADS-A (<8 on a scale 0-21 with high numbers indicating increased anxiety)
Self-rated quality-of-life determined by Research ANd Development-36 (RAND-36) | 10, 20 and 50 weeks after randomisation
  RAND-36: 0-100 with high numbers indicating better quality-of-life
Self-rated cardiac anxiety determined by Cardiac Anxiety Questionnaire (CAQ) | 10, 20 and 50 weeks after randomisation
  CAQ: 0-72 with high numbers indicating increased cardiac anxiety
Self-rated post-traumatic symptoms determined by Impact of Event Scale-6 (IES-6) | 10, 20 and 50 weeks after randomisation
  IES-6: 0-30 with high numbers indicating increased post-traumatic symptoms
Sick leave | 10, 20 and 50 weeks after randomisation
  Self-reported total number of days
Health-care visits | 10, 20 and 50 weeks after randomisation
  Self-reported total number of visits
Cortisol in hair | 10 weeks after randomisation
  Hair cortisol will be determined by RIA-technique in pg/mg
Physiological recovery after stress determined by Heart Rate Variability (HRV) | 10 weeks after randomisation
  HRV will be measured by time and frequency domains and by non-linear methods
Physiological recovery after stress determined by salivary cortisol | 10 weeks after randomisation
  Salivary cortisol will be determined by RIA-technique in pg/mg

CONTACTS AND LOCATIONS:
Locations (1):
- Södersjukhuset, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rondung E, Humphries SM, Olsson EMG, Sundelin R, Norlund F, Held C, Spaak J, Tornvall P, Lynga P. Reducing stress and anxiety in patients with myocardial infarction with non-obstructive coronary arteries or Takotsubo syndrome: A non-randomized feasibility study. Internet Interv. 2022 Jul 21;29:100562. doi: 10.1016/j.invent.2022.100562. eCollection 2022 Sep. PMID 35910688
- [Derived] Olsson EMG, Norlund F, Rondung E, Humphries SM, Held C, Lynga P, Spaak J, Sundin O, Sundelin R, Leissner P, Kovamees L, Tornvall P. The e-mental health treatment in Stockholm myocardial infarction with non-obstructive coronaries or Takotsubo syndrome study (E-SMINC): a study protocol for a randomised controlled trial. Trials. 2022 Jul 26;23(1):597. doi: 10.1186/s13063-022-06530-3. PMID 35883115

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-08-24): https://cdn.clinicaltrials.gov/large-docs/34/NCT04178434/Prot_SAP_002.pdf